CLINICAL TRIAL: NCT02870543
Title: Efficacy of Phytolacca Decandra and Melissa Officinalis in Children With Nocturnal Bruxism: a Controlled and Randomized Clinical Trial
Brief Title: Efficacy of Phytolacca Decandra and Melissa Officinalis in Children With Nocturnal Bruxism
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Cláudia Maria Tavares da Silva, Ph.D student, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 37302414.2.0000.5257
Record Dates: First submitted 2016-07-28; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Nocturnal Bruxism
Keywords: Bruxism; Sleep bruxism; Sleep related bruxism; Homeopathy
MeSH Terms: conditions — Sleep Bruxism; Bruxism | interventions — Homeopathy; lemon balm leaf extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Phytolacca decandra; Drug: Melissa officinalis; Drug: Phyt.decandra + Melissa offic.
- Phytolacca decandra (Active Comparator): The Phytolacca decandra with 12CH dosage will be administered (one drop per age of the child) once a day during 30 days.
  Interventions: Drug: Melissa officinalis; Drug: Phyt.decandra + Melissa offic.
- Melissa officinalis (Active Comparator): The Melissa officinalis with 12CH dosage will be administered (one drop per age of the child) once a day during 30 days.
  Interventions: Drug: Phytolacca decandra; Drug: Phyt.decandra + Melissa offic.
- Phyt.decandra + Melissa offic. (Experimental): The combination of Phytolacca decandra with Melissa offcicinalis with 12CH dosage will be administered (one drop per age of the child) once a day during 30 days.
  Interventions: Drug: Phytolacca decandra; Drug: Melissa officinalis

INTERVENTIONS:
Drug: Phytolacca decandra — Treatment of bruxism
  Other Names: homeopathic medicine
  Arms: Melissa officinalis; Phyt.decandra + Melissa offic.; Placebo
Drug: Melissa officinalis — Treatment of bruxism
  Other Names: homeopathic medicine
  Arms: Phyt.decandra + Melissa offic.; Phytolacca decandra; Placebo
Drug: Phyt.decandra + Melissa offic. — Treatment of bruxism
  Other Names: homeopathic medicine complex
  Arms: Melissa officinalis; Phytolacca decandra; Placebo

SUMMARY:
This study aims to evaluate, through a crossover, controlled, double-blind and randomized clinical trial, the efficacy of Phytolacca decandra in association or not with Melissa officinalis in the treatment of children with nocturnal bruxism. Children from 3 to 12 years old with nocturnal bruxism will be randomly allocated into different groups of treatment stage as follows: (1) placebo; (2) Phytolacca decandra; (3) Melissa officinalis; (4) Phytolacca decandra associated with Melissa officinalis. All children will participate to each clinical stage, with a period of 14 days of whashout. Children and the principal investigator will be masked to treatment. The efficacy will be evaluated through parents report about the absence of tooth clenching or grinding by children and electromiography exams. The secondary outcomes that will be evaluated are: trait anxiety and quality of life related to oral health.

DETAILED DESCRIPTION:
This is a randomized, double-blind, crossover, placebo-controlled study in which children aged 3 to12 years old with nocturnal bruxism will be randomly allocated into different phases of the study, according to treatment step: (1) placebo; (2) Phytolacca decandra; (3) Melissa officinalis; (4) Phytolacca decandra associated with Melissa officinalis. This study will be enrolled in Dental clinic of the Pediatric Dentistry department of Dental School, in Federal University of Rio de Janeiro (UFRJ), from September 2014 to July 2017. All children will participate of each clinical stages, with a washout interval of 14 days between the phases. Children and the principal investigator will be masked to treatment.

After anamnesis, extra and intraoral clinical examination will be conducted at the beginning of the study, by a single trained and calibrated examiner (the researcher responsible for the study). Thus, facial symmetry, temporomandibular joints and masticatory muscle activity should be observed. For the evaluation of the residual effect of bruxism in the muscles (masseter and temporalis) of the masticatory system, electromyography exams will be performed.

For intra-oral clinical examination, patients will be positioned comfortably in a dental chair and the exam will be conducted with the aid of artificial light from dental reflector mirror plane, exploratory probe and cotton tweezers. Data from each patient will also be recorded in the dental records by a previously trained annotator. The presence of clinical signs related to the presence of bruxism, such as the presence of dental enamel wear and microfractures facets will also be evaluated.

The Brazilian version of ECOHIS (B-ECOHIS) will be used to assess the quality of life for the selected children with 0-7 years old. This instrument will be applied before and after each phase of the study. And, the Brazilian version of "Child Perceptions Questionnaire" (CPQ) 8-10 and 11-14, will also be used to assess the physical and psychosocial impact of nocturnal bruxism in children and adolescents in the study.

The child's anxiety will be observed by means of a rating scale of trait anxiety in children. This scale will also be applied before and after each phase of the study.

All medicines, including placebo, will be placed in identical amber glass vials, which will be labeled / encoded (A, B, C, D) and distributed ramdonly to children/parents, in accordance with the phases of the study.

In every return, parents / guardians must give back the bottle used in the period to be verified the residual volume. Thus, the intake of the medicine will be properly evaluated.

The subjects will be distributed within the treatment phases of the study in accordance with the following medications:• Phase 1 - Placebo; • Phase 2 - Use isolated of Phytolacca decandra 12CH; • Phase 3 - Use isolated of Melissa officinalis 12CH; • Phase 4 - Combined use of Phytolacca decandra 12CH and Melissa officinalis 12CH.

Each drug, including placebo, will be formulated in Homeopathy Pharmacy, Faculty of Pharmacy, UFRJ. They will be administered for a period of 30 days with a washout interval of 14 days between phases.

All test solutions will be packed in amber glass 30 ml with dropper and will be prepared at the same time and under the same laboratory conditions. Supervision of all pharmaceutical manipulation will be under the technical responsibility of at least one homeopathic pharmaceutic.

Administration of the test medicines (solutions) will be made once a day, with the following dosage: 01 drops of solution per age of the individual.

Patients and their caregivers must be informed that all products involving oral care (toothpastes and mouthwashes) interfere with the absorption of homeopathic medicine, so the 15-minute interval should be preserved between the drug intake and self-care mouth of each individual. It is emphasized that the use of the drug, quantity, time and frequency will be informed through a written prescription.

The parents and/ or guardians will be responsible for helping monitoring the efficacy of the treatments. At the first visit, they will receive a notebook that will serve as a sleep diary. This instrument will be used for parents and / or guardians to describe their self-perception of the sleep routine of their children.

In this appointment the parents and / or guardians will receive the researcher's instructions about the completion of the daily diary. Thus, it will serve later as the child's primary information before starting the use of medicines. This routine should be maintained throughout the period of treatment, and in the resting phase (wash out), serving as a home mirror, reflecting the effects presented by the child during the study period.

The frequency of nocturnal bruxism will be assessed using a Visual Analogue Scale. This scale will be applied to parents and / or guardians in the first appointment to obtain the frequency of bruxism of each child at the baseline. Also, it will be reapplied during all phases for monitoring the clenching and grinding of the teeth.

A multiple logistic regression model will be applied to investigate the difference between treatments.

ELIGIBILITY:
Inclusion criteria:

* Children with good general health; children aged 03-12 years old; children with nocturnal bruxism reported by their parents/guardians.

Exclusion criteria:

* Children with special needs (frame psychological, psychiatric and neurological disorders or any systemic commitments)
* Children with carious lesions in dentin
* Children with orthodontic appliances
* Children with dental anomalies
* Children with dental erosions
* Children with the following malocclusions: Class II and III of Angle, crossbite and open bite
* Children that will be in any medication that modify the salivary flow and / or cause alteration of the central nervous system.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of efficacy of Phytolacca decandra in association or not with Melissa officinalis in comparison of placebo in arresting nocturnal bruxism, by the use of a visual analog scale | During the period of treatments and washout : 168 days
  Parents / guardians will be asked to schedule a graduated visual analog scale from 0 to 10 to determine bruxism level (absence or not of tooth clenching or grinding) of your child during the 30 days of each medicine usage and also during the washout period.
Evaluation of the efficacy of Phytolacca decandra in association or not with Melissa officinalis in comparison of placebo in arresting nocturnal bruxism, by the electromiography analysis | Before to start all treatments (baseline) and after each treatment (every 30 days) up to 168 days
  All children will be submitted to eletromiography analysys to measure the masseter and temporalis muscles forces before and after each tretament stage.

SECONDARY OUTCOMES:
Identify changes in the quality of life children with bruxism before and after treatments by the use of B-ECOHIS and PCP-Q questionaries | Before to start all treatments (baseline) and after each treatment (every 30 days) up to 168 days
  Parents / guardians will answer questionnaires to determine their children' quality of life related to oral health before and after each stage of the study.

OTHER OUTCOMES:
Identify changes in the trait anxiety of children with bruxism before and after treatments by the use of the Brazilian validated version of the Trait-anxiety Scale | Before to start all treatments (baseline) and after each treatment (every 30 days) up to 168 days
  Parents/guardians will answer the questionnaire (the Brazilian validated version of the Trait-anxiety Scale) to determine their children trait anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea G. Antonio, Adjunct Professor, Study Chair — Universidade Federal do Rio de Janeiro; Lucianne Cople Maia, Full Professor, Study Director — Universidade Federal do Rio de Janeiro; Cláudia Tavares, Ph.D student, Principal Investigator — Universidade Federal do Rio de Janeiro

IPD SHARING:
Plan to Share IPD: Undecided